CLINICAL TRIAL: NCT05626556
Title: A Technology-based Intervention to Support Older Adults in Living Independently: Protocol for a Cross-national Feasibility Pilot
Brief Title: A Technology-based Intervention to Support Older Adults in Living Independently
Acronym: SAVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_005_2022
Record Dates: First submitted 2022-11-11; First posted 2022-11-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-11

CONDITIONS: Older People; Frailty
Keywords: technology-based intervention; older adults; active ageing
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- older adults (Experimental): Older adults with mild to moderate chronic illness
  Interventions: Other: SAVE system

INTERVENTIONS:
Other: SAVE system — The SAVE system will be implemented in end users' homes. Flood sensors will be installed in the bathroom and kitchen, presence sensors in the living room and bedroom, and the contact sensor will be installed at the entrance door. For the best user experience, the installation of the required software (for the sensors kit and the smartwatch) was done on the users' own smartphones. Thus, at the end of the installation, users will have the Aqara Home System in their homes (5 sensors and a sensor hub), a Samsung smartwatch and a SAVE Sensors Adapter, all of which are connected to a router with unlimited internet access.

SUMMARY:
The general objective of this study is to test the usability and efficiency of the SAVE prototype, a technology-based support for enabling older adults to keep their independent and active lives in their homes and maintain their social relationships for as long as possible.

DETAILED DESCRIPTION:
The SAVE system aims to offer technology-based support to older adults for staying in their familiar surroundings for as long as possible, while feeling safe and optimally cared for. The SAVE technology has been designed and developed according to the approach of the User Centered Design (UCD), which involves multiple interactions with users to under-stand their needs and preferences and to involve them in the design process for creating a truly useful and appreciated technological product. Secondarily, it supports informal caregivers, like relatives, in providing optimal care for their loved ones, while maintaining their professional and private life. The general objective of this study is to test the usability and efficiency of the SAVE prototype for enabling older adults to keep their independent and active lives in their homes and maintain their social relationships for as long as possible. The study involves the use of the SAVE platform for a total of 21 consecutive days.The study involves the use of a mixed-methods approach, in which both qualitative (open questions) and quantitative (standardized tests) data will be collected, and three different measurements (T0, T1, T2) will be made during the period of use of the system. The data collection card will therefore be divided into two different sections, which correspond to the three different moments of detection: 1) at time 0, that is, before the start of the experi-mentation (T0); 2) at time 1, after 10 days, i.e. at the midterm of the trial (T1), and 3) at time 2, after 21 days, i.e., at the end of the trial (T2). The log data of the usage of the SAVE sys-tem be the primary, secondary, and tertiary users will be continuously stored over the 21 days test period.

ELIGIBILITY:
Inclusion Criteria:

* Mini Mental State Evaluation (MMSE) between 21 and 24
* Healthy or mild to moderate chronic illness or musculoskeletal disease
* Feel physically fit to participate in the study

Exclusion Criteria:

* Participants suffer from severe chronic disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Usability | Change from baseline SUS at 21 days from the start of the intervention
  This outcome will be measured through the System Usability Scale (SUS). It consists of a 10-item questionnaire with five response options for respondents from 'Strongly agree' to 'Strongly disagree'.
Acceptance | Change from baseline UEQ at 21 days from the start of the intervention
  This outcome will be measured through the the User Experience Questionnaire (UEQ). The UEQ is a semantic differential with 26 items. The scales of the questionnaire cover a comprehensive impression of user experience. Items are scored on a 7-point Likert scale and range from full agreement with the negative term (-3) to the full agreement with the positive term (+3). Half of the items start with the positive term, the rest with the negative term. Higher sum scores indicate more positive evaluation.

SECONDARY OUTCOMES:
Cognitive impairment | at baseline, at 10 days from the start of the intervention and at 21 days from the start of the intervention
  This outcome will be measured by Mini-Mental State Examination (MMSE). It is a neuropsychological test for the evaluation of disorders of intellectual efficiency and the presence of cognitive impairment. The total score is between a minimum of 0 and a maximum of 30 points. A score of 26 to 30 is an indication of cognitive normality. The score will be adjusted with the coefficient for age and schooling.
Autonomy in walking | at baseline, at 10 days from the start of the intervention and at 21 days from the start of the intervention
  This outcome will be measured by the Ambulation Category (FAC). It is a scale that evaluates the ability to autonomy in walking. The ambulatory capacity is evaluated with a score ranging from 0 to 5, where 0 indicates total dependence and 5 complete autonomy.
Functional status | at baseline, at 10 days from the start of the intervention and at 21 days from the start of the intervention
  This outcome will be measured by the Barthel Index. The individual is scored in a number of areas depending upon independence of performance. Total scores range from 0 (complete dependence) to 100 (complete independence).
State of health | at baseline, at 10 days from the start of the intervention and at 21 days from the start of the intervention
  This outcome will be measured by the SF-12v2 ™ Health Survey. It is a widely used instrument, and is a 12-element sub-set of the SF-36v2™. This is a generic assessment of the health-related quality of life from the patient's perspective. The mean score is set to 50. Scores >50 indicate better physical or mental health than the mean. Scores <50 indicate worse physical or mental health than the mean.

CONTACTS AND LOCATIONS:
Locations (3):
- Országos Orvosi Rehabilitációs Intézet, Szanatórium, Budapest, Hungary
- IRCCS INRCA Hospital, Ancona, Italy
- Transilvania University of Brașov, Brasov, Romania

REFERENCES:
- [Derived] Stara V, Rampioni M, Mosoi AA, Kristaly DM, Moraru SA, Paciaroni L, Paolini S, Raccichini A, Felici E, Rossi L, Vizitiu C, Nistorescu A, Marin M, Tonay G, Toth A, Pilissy T, Fazekas G. A Technology-Based Intervention to Support Older Adults in Living Independently: Protocol for a Cross-National Feasibility Pilot. Int J Environ Res Public Health. 2022 Dec 10;19(24):16604. doi: 10.3390/ijerph192416604. PMID 36554485